CLINICAL TRIAL: NCT00088660
Title: A Phase III Randomized, Controlled Study to Evaluate the Safety and Efficacy of PANVAC™-VF in Combination With GM-CSF Versus Best Supportive Care or Palliative Chemotherapy in Patients With Metastatic (Stage IV) Adenocarcinoma of the Pancreas Who Have Failed a Gemcitabine-Containing Chemotherapy Regimen
Brief Title: PANVAC™-VF Vaccine for the Treatment of Metastatic Pancreatic Cancer After Failing a Gemcitabine-Containing Regimen
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Therion Biologics Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBC-PAN-003
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2006-02

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Biological: PANVAC™-VF

SUMMARY:
The objectives of this multi-center, randomized, controlled trial are to evaluate the safety and efficacy of PANVAC-VF in combination with Granulocyte-macrophage colony-stimulating factor (GM-CSF) versus best supportive care or palliative chemotherapy.

DETAILED DESCRIPTION:
PANVAC-VF is an investigational cancer vaccine. The vaccine is based on the theory that the body can be taught to fight cancer by directing the immune system to attack specific targets found on cancer cells. These targets are called Tumor Associated Antigens, or TAA's. This trial will help determine if this vaccine can help fight cancer.

All patients will be required to sign an informed consent prior to the performance of any study-related procedures. Patients will be screened for eligibility within 14 days prior to their anticipated treatment start date (Day 0). Patients who meet all inclusion and exclusion criteria will be centrally randomized into the study and will receive a unique patient identification number and a treatment assignment. The ratio of active treatment to control is 1:1 (PANVAC-VF: best supportive care or palliative chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age who have been vaccinated against smallpox;
* Histologically confirmed diagnosis of adenocarcinoma of the pancreas;
* Patient has metastatic (Stage IV) disease;
* ECOG performance status 0-1;
* Failed a gemcitabine-containing chemotherapeutic regimen within 3 months of study entry.

Exclusion Criteria:

* Prior or concurrent immunotherapy for cancer;
* Radiation therapy within 28 days prior to registration;
* Systemic corticosteroid therapy (except inhaled or topical steroids) within 28 days of registration;
* Significant cardiovascular abnormalities or diseases;
* Known positive for HIV, hepatitis B and/or C;
* Evidence of immunodeficiency or immune suppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - University of South Alabama/ Cancer Research Institute, Mobile, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Chao Family Comprehensice Cancer Center, Orange, California
  - Desert Hematology Oncology Medical Group, Inc, Rancho Mirage, California
  - Scripps Cancer Center, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - Greeley Medical Clinic, Greeley, Colorado
  - Loveland Hematology Oncology, Loveland, Colorado
  - Norwalk Hospital/ Whittingham Cancer Center, Norwalk, Connecticut
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Washington Hospital Cancer Center, Washington D.C., District of Columbia
  - Jupiter Medical Center, Jupiter, Florida
  - VA Medical Center, Miami, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Sylvester Cancer Center, Miami, Florida
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Carle Cancer Center, Urbana, Illinois
  - Oncology Associates, Cedar Rapids, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - Jayne Gurtler, MD and Laura Brinz, MD APMC, Metairie, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Franklin Square Hospital, Baltimore, Maryland
  - Tufts-New England Medical Center, The Neeley Center for Clinical Research, Boston, Massachusetts
  - Josephine Ford Cancer Center, Detroit, Michigan
  - Kansas City Cancer Center, Kansas City, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Winthrop Oncology/Hematology Division, Mineola, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Dayton Oncology Hematology, Kettering, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Temple University Cancer Center, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Cancer Care, Fort Worth, Texas
  - Dr. H. Alejandro Preti, F.A.C.P., Houston, Texas
  - Elkins Pancreas Center, Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Cancer Care, Weatherford, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Medical Consultants Ltd., Milwaukee, Wisconsin